CLINICAL TRIAL: NCT03225378
Title: Changes in Pulse Pressure Variations Induced by Passive Leg Raising Test to Predict Fluid Responsiveness in ICU
Brief Title: Changes in PPV Induced by PLR Test to Predict Fluid Responsiveness in ICU
Acronym: VPP-ImPRoVE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Arras (Other)
Responsible Party: Sponsor
Other Study IDs: 2017_01
Record Dates: First submitted 2017-07-20; First posted 2017-07-21 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Acute Circulatory Failure
Keywords: Fluid responsiveness; Passive leg raising; Pulse pressure variation
MeSH Terms: conditions — Shock | interventions — Crystalloid Solutions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute circulatory failure: Mechanically ventilated patients displaying acute circulatory failure in whom the physician decides to perform a fluid challenge (fluid loading of 500 mL of crystalloid solution) and a passive leg raising test to predict fluid responsiveness.
  Interventions: Other: Fluid loading of 500 mL of crystalloid solution; Other: Passive Leg Raising test

INTERVENTIONS:
Other: Fluid loading of 500 mL of crystalloid solution — Infusion of 500 mL of crystalloid solution in less than 15 minutes
Other: Passive Leg Raising test — This intervention is done before the fluid loading in order to predict fluid responsiveness.

SUMMARY:
The passive leg raising (PLR) test is a reversible preload challenge of around 300 mL of blood that can be repeated as frequently as required without infusing a drop of fluid. Two recent meta-analyses of many studies have confirmed the reliability of the PLR test to predict fluid responsiveness in patients with acute circulatory failure. Nevertheless, the effects of the PLR must be assessed by the direct measurement of cardiac output since changes in arterial pressure do not allow the assessment of the PLR hemodynamic effects with reliability. Moreover, cardiac output must be measured continuously and in real time.

In clinical practice, cardiac output measurement can be difficult for different reasons such as the unavailability of the echocardiography machine, or the absence of any continuous cardiac output monitoring technique at the time of acute circulatory failure occurrence.

Recently, it was shown that the decrease in pulse pressure variation (PPV) induced by the mini-fluid challenge (100 mL of colloid solution infused in 1 min) was able to predict fluid responsiveness with reliability in patients ventilated with low tidal volume (<8 mL/kg of ideal body weight).

Therefore, the investigators hypothesize that the changes in PPV induced by PLR test could be able to predict fluid responsiveness with reliability in mechanically ventilated patients with acute circulatory failure.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated patients
* Patients in whom the physician decides to perform a fluid challenge based on the presence of one of the following criteria:

  (1) systolic arterial pressure <90 mmHg, mean arterial pressure <65 mmHg, or the need for vasopressor infusion; (2) skin mottling; (3) urine output <0.5 mL/Kg/h for more than or equal to 2 hours; (4) lactate concentrations > 2 mmol/L
* Patients in whom the physician decides to perform a PLR test to predict fluid responsiveness
* Arterial catheter should be in place for invasive monitoring of arterial pressure and PPV

Non inclusion Criteria:

* Age <18 yrs
* Pregnancy
* Moribund patients
* Risk of fluid loading induced pulmonary edema
* Cardiac arrhythmias
* Contraindication to perform PLR (intracranial hypertension, pelvic fractures)

Exclusion Criteria :

* Changes in vasopressor and sedation agents dosages during the protocol
* Changes in ventilatory parameters during the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients displaying acute circulatory failure signs in whom the physician decides to perform a fluid challenge and a PLR test to predict fluid responsiveness.
Sampling Method: Non-Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Increase in cardiac output in all mechanically ventilated patients | Cardiac output will be measured immediately after the end of the volume expansion
  The primary endpoint is the increase in cardiac output of more than or equal to 15% after 500 mL of volume expansion. All included patients are concerned by the primary outcome.

SECONDARY OUTCOMES:
Increase in cardiac output in mechanically ventilated patients with spontaneous breathing activities | Cardiac output will be measured immediately after the end of the volume expansion
  The secondary endpoint is the increase in cardiac output of more than or equal to 15% after 500 mL of volume expansion. Only patients with spontaneous breathing activities are concerned by this secondary outcome.
Increase in cardiac output in mechanically ventilated patients with low tidal ventilation and/or low respiratory compliance | Cardiac output will be measured immediately after the end of the volume expansion
  The secondary endpoint is the increase in cardiac output of more than or equal to 15% after 500 mL of volume expansion. Only patients with low tidal ventilation (<8mL/kg of ideal body weight) and/or low respiratory compliance (<30mL/cmH2O) are concerned by this secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jihad MALLAT, MD, Principal Investigator — Centre Hospitalier Arras
Locations (12):
- France (12):
  - CHU d'Amiens - Réanimation Cardio-Thoracique-Vasculaire, Amiens
  - CHU d'Amiens - Réanimation chirurgicale, Amiens
  - Centre Hospitalier d'Arras, Arras
  - Centre Hospitalier de Béthune, Béthune
  - CH Boulogne-sur-mer, Boulogne-sur-Mer
  - CHU de Caen, Caen
  - Centre Hospitalier de Cambrai, Cambrai
  - CHU de Dijon, Dijon
  - Centre Hospitalier de Lens - Anesthésie-Réanimation, Lens
  - Centre Hospitalier de Lens - Réanimation, Lens
  - CHRU de Lille - Réanimation Médicale, Lille
  - CHU de Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Monnet X, Marik P, Teboul JL. Passive leg raising for predicting fluid responsiveness: a systematic review and meta-analysis. Intensive Care Med. 2016 Dec;42(12):1935-1947. doi: 10.1007/s00134-015-4134-1. Epub 2016 Jan 29. PMID 26825952
- [Result] Cherpanath TG, Hirsch A, Geerts BF, Lagrand WK, Leeflang MM, Schultz MJ, Groeneveld AB. Predicting Fluid Responsiveness by Passive Leg Raising: A Systematic Review and Meta-Analysis of 23 Clinical Trials. Crit Care Med. 2016 May;44(5):981-91. doi: 10.1097/CCM.0000000000001556. PMID 26741579
- [Result] Mallat J, Meddour M, Durville E, Lemyze M, Pepy F, Temime J, Vangrunderbeeck N, Tronchon L, Thevenin D, Tavernier B. Decrease in pulse pressure and stroke volume variations after mini-fluid challenge accurately predicts fluid responsivenessdagger. Br J Anaesth. 2015 Sep;115(3):449-56. doi: 10.1093/bja/aev222. Epub 2015 Jul 6. PMID 26152341
- [Derived] Mallat J, Abou-Arab O, Lemyze M, Saleh D, Guinot PG, Fischer MO. Changes in central venous-to-arterial PCO2 difference and central venous oxygen saturation as markers to define fluid responsiveness in critically ill patients: a pot-hoc analysis of a multi-center prospective study. Crit Care. 2024 Nov 8;28(1):360. doi: 10.1186/s13054-024-05156-y. PMID 39516883
- [Derived] Mallat J, Lemyze M, Fischer MO. Passive leg raising test induced changes in plethysmographic variability index to assess fluid responsiveness in critically ill mechanically ventilated patients with acute circulatory failure. J Crit Care. 2024 Feb;79:154449. doi: 10.1016/j.jcrc.2023.154449. Epub 2023 Oct 17. PMID 37857068
- [Derived] Mallat J, Fischer MO, Granier M, Vinsonneau C, Jonard M, Mahjoub Y, Baghdadi FA, Preau S, Poher F, Rebet O, Bouhemad B, Lemyze M, Marzouk M, Besnier E, Hamed F, Rahman N, Abou-Arab O, Guinot PG. Passive leg raising-induced changes in pulse pressure variation to assess fluid responsiveness in mechanically ventilated patients: a multicentre prospective observational study. Br J Anaesth. 2022 Sep;129(3):308-316. doi: 10.1016/j.bja.2022.04.031. Epub 2022 Jul 14. PMID 35842352